CLINICAL TRIAL: NCT01142050
Title: A Open Labeled and Self Controlled, Safety/Efficacy Assessed Pilot Study on Transplantation Therapy Using Bone Marrow Mesenchymal Stem Cells for Insulin Resistance of Type 2 Diabetes Mellitus
Brief Title: Stem Cell Therapy for Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cellonis Biotechnology Co. Ltd. (Industry)
Responsible Party: Cellonis Biotechnology Co. Ltd., others
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cellonis-CR-2.3
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: stem cells;; diabetes mellitus;; treatment.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Biological: mesenchymal stem cells — 1.1st transplantation: after finishing all required examines according to protocol in Day 0, ABM-MSCs are transplanted through pancreas artery percutaneously; 2. 2nd transplantation: after finishing all required examines in Day 7±1, BM-MSCs are transplanted intravenously; 3. 3rd transplantation: after finishing all required examines in Day 14±2, BM-MSCs are transplanted intravenously.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety in the treatment of Insulin Resistance of Type 2 Diabetes Mellitus with Bone Marrow Mesenchymal Stem Cells.

DETAILED DESCRIPTION:
* To evaluate the feasibility and safety of transplantation treatment using umbilical cord mesenchymal stem cells in patients with type 2 diabetes mellitus undergoing insulin injection treatments.
* To assess efficacy of transplantation treatment using umbilical cord mesenchymal stem cells in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Free will taking part in the study and ability to provide written informed consent;
2. Type 2 diabetes mellitus (as guideline WHO, 1999);
3. Age 18-75 years old，Male/Female;
4. 19≤Body mass index (BMI)≤30㎏/㎡;
5. Fast blood glucose (FBG)≥7.0 mmol/L, and HbAc1≥7％;
6. Intravenous insulin tolerance test（ITT）indicate patient being insulin resistance;
7. Not pregnant or nursing;
8. Negative pregnancy test;
9. Fertile patients will use effective contraception.

Exclusion Criteria:

1. Severe concurrent medical condition (e.g., serious heart disease, lung disease, or hematopoietic dysfunction, or liver dysfunction, or kidney dysfunction);
2. Active infection requiring treatment;
3. Unexplained febrile illness;
4. Known immunosuppressive disease, e.g. HIV infection, or hepatitis B or C infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
ITT; insulin dosage; Hemoglobin A1c; Fast blood glucose (FBG) and Postmeal blood glucose (PBG); C-peptide levels; Serum Insulin levels; | one year
  1. Insulin resistance index indicated by ITT change compared with baseline.
  2. Rate of reducing exogenous insulin requirement and OGLD dosage compared with baseline.
  3. Hemoglobin A1c.
  4. Fast blood glucose (FBG) and Postmeal blood glucose (PBG).
  5. C-peptide levels.
  6. Serum Insulin levels.

SECONDARY OUTCOMES:
Serious adverse event frequency and severity | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Police General Hospital, P.R. China, Beijing, China